CLINICAL TRIAL: NCT04010110
Title: Hydroxychloroquine Dosing and Toxicity in Ophthalmology Clinics
Status: Completed | Type: Observational
Sponsor: The Eye Center and The Eye Foundation for Research in Ophthalmology (Other)
Collaborators: King Khalid University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TEC 2017-003
Record Dates: First submitted 2019-07-02; First posted 2019-07-08 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Hydroxychloroquine Toxic Retinopathy
Keywords: Hydroxychloroquine; Toxic retinopathy; Hydroxychloroquine screening
MeSH Terms: interventions — Visual Fields

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients on hydroxychloroquine: A data collection sheet was used to collect patient's information. All patients underwent a complete ophthalmic examination including assessment of visual acuity, anterior segment examination looking for corneal verticillata and a dilated fundus examination looking for retinal pigment epithelium (RPE) depigmentation either in a para-foveal or extra-macular distribution within the retina. Ancillary tests were done which included: visual field testing (10-2), spectral domain ocular coherence tomography (SDOCT). Fundus auto-fluorescence and mf-ERG were done if further ancillary testing was needed in doubtful cases or to confirm findings.
  Interventions: Diagnostic Test: visual field testing (10-2), spectral domain ocular coherence tomography and Fundus auto-fluorescence

INTERVENTIONS:
Diagnostic Test: visual field testing (10-2), spectral domain ocular coherence tomography and Fundus auto-fluorescence — The diagnosis of toxic retinopathy was based on the positivity of at least two objective tests to confirm the subjective findings. The presence or absence of toxicity was recorded.

SUMMARY:
This study assesses the ocular toxicity in patients on high dose hydroxychloroquine (HCQ) as per the latest guidelines of the American Academy of Ophthalmology (AAO).

DETAILED DESCRIPTION:
Hydroxychloroquine (HCQ) is an anti-malarial drug that is used to treat a variety of autoimmune diseases, such as rheumatoid arthritis and systemic lupus erythematosus, juvenile idiopathic arthritis and Sjogren's syndrome. Hydroxychloroquine is a less toxic metabolite of chloroquine. There is an ongoing increase in the number of patients who are using HCQ for prolonged duration because of the expanding indications and the relatively safe systemic profile.

Hydroxychloroquine can cause variable ocular adverse effects including corneal deposits, posterior sub-capsular cataract, ciliary body dysfunction and toxic retinopathy. Toxic retinopathy caused by HCQ has been recognized for many years. Patients with toxic retinopathy usually complain of blurry vision. The classical clinical picture of HCQ toxic retinopathy is a bilateral bull's-eye maculopathy, which is caused by a ring of parafoveal RPE depigmentation that spares the fovea. The exact mechanism responsible for the development of this pattern is not fully understood, however, it is believed that the primary damage is in the photoreceptors and outer nuclear layer leading to secondary disruption of the RPE.

ELIGIBILITY:
Inclusion Criteria:

* Patients on hydroxychloroquine therapy who came for their ophthalmology screening appointment irrespective of the duration of use of the medication.

Exclusion Criteria:

* Patients who have stopped their hydroxychloroquine medication.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending the ophthalmology clinics at King Khalid University Hospital and The Eye Center in Riyadh, Saudi Arabia.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by clinical signs and ancillary tests | 2 years
  A data collection sheet used to collect patient's information regarding the dose per body weight and duration of hydroxychloroquineuse and any risk factors associated with the use of the medication as per the latest AAO guidelines for hydroxychloroquine screening.
  Complete ophthalmic examination including assessment of visual acuity, anterior segment examination looking for corneal verticillata and a dilated fundus examination looking for retinal pigment epithelium (RPE) depigmentation either in a para-foveal or extra-macular distribution within the retina. Ancillary tests including visual field (10-2) testing, spectral domain ocular coherence tomography (SDOCT) fundus auto-fluorescence and multifocal Electroretinogram (ERG).

CONTACTS AND LOCATIONS:
Locations (1):
- The Eye Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No